CLINICAL TRIAL: NCT02158013
Title: Treatment Of Chronic Anal Fissure (TOCA): a Randomized Clinical Trial on Levorag® Emulgel Versus Diltiazem Gel 2%
Brief Title: Treatment Of Chronic Anal Fissure
Acronym: TOCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Sacomed (Other)
Responsible Party: Principal Investigator, Peter-Martin Krarup, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-6-2014-020
Record Dates: First submitted 2014-06-05; First posted 2014-06-06 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Levorag; Diltiazem

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diltiazem, calcium channel blocker (Active Comparator): Diltiazem gel 2% applied twice daily for 8 weeks
  Interventions: Drug: Diltiazem
- Levorag, Hibiscus plant extract (Experimental): Levorag Emulgel applied twice daily for 8 weeks
  Interventions: Other: Levorag Emulgel

INTERVENTIONS:
Other: Levorag Emulgel
  Other Names: Myoxinol; Carboxymethyl glucan
  Arms: Levorag, Hibiscus plant extract
Drug: Diltiazem
  Arms: Diltiazem, calcium channel blocker

SUMMARY:
The purpose of this study is to investigate the effect of Levorag Emulgel compared with diltiazem gel on the healing of chronic anal fissures.

DETAILED DESCRIPTION:
Anal fissure is an ulcer-like, longitudinal tear in the anal canal, most commonly located in the dorsal or ventral midline, and distal to the dentate line. Anal fissures constitute a common medical problem that affects sexes equally. The initiation of the fissure is most likely caused by the passage of hard stools that traumatizes the anal canal. Patients suffer from anal pain lasting up to several hours after defecation and rectal bleeding.3 Most acute anal fissures heal spontaneously, but a proportion progress into chronic fissures with symptoms beyond 8-12 weeks. There is no strict definition of a chronic anal fissure, but previously the presence of two of the following three symptoms has been used:

1. Pain after defecation lasting for more than three months;
2. presence of a sentinel anal tag; and
3. Exposure of the horizontal fibres of the internal anal sphincter. The severe pain may be caused by a hypertonic contraction of the internal anal sphincter leading to ischemia. Treatment strategies have therefore aimed to relieve this hypertonia by surgical and non-operative approaches. Primary therapy is initiated with ointments such as Diltiazem and glyceryltrinitrat gels.

A novel approach is the Levorag® Emulgel, an ointment classified as Medical Device class 1. According to the manufacturer (THD SpA, Italy) the effect of Levorag® Emulgel is mediated through the effects of myoxinol, a plant extract from the Hibiscus plant with a botox-like effects on the anal sphincter and carboxymethyl glucan, a natural yeast polysaccharide with immune stimulating properties. The effect of the widely used Diltiazem gel, is mediated through diltiazem hydrochloride, a calcium channel blocker that decreases the anal sphincter pressure.

This is an interventional, randomized clinical trial including adult patients with chronic anal fissures referred directly to the Digestive Disease Center, Bispebjerg Hospital, University of Copenhagen, or referred to a private surgical practice in Copenhagen. Patients are randomized to 1) Diltiazem gel 2%, one application twice daily for 8 weeks, or 2) Levorag® Emulgel, one application twice daily for 8 weeks. In addition to the allocated treatment, all patients will be kept on standard care for anal fissure, including high-fibre diet proper hydration and laxatives.

The primary endpoint is the rate of complete healing after 12 weeks. Secondary endpoints are complete healing after 8 weeks, incidence of adverse effects and efficacy on pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. Danish citizens, age ≥ 18 years
2. Presence of a midline anal fissure, dorsal or ventral
3. Pain during and after defecation lasting for more than 8 weeks
4. Presence of a sentinel anal tag or hypertrophic papilla
5. Exposure of the horizontal fibres of the internal anal sphincter

1-3 has to be fulfilled for inclusion. Additionally 4 AND/OR 5 has to be present

Exclusion Criteria:

1. Inflammatory bowel disease, known venereal disease, immunodeficiency disease
2. Anal/perianal abscess
3. Anal or rectal surgery within 12 weeks
4. Pregnancy or breastfeeding females
5. History of migraine or chronic headache requiring treatment with analgetics
6. Any cardiovascular or cerebrovascular disease
7. Current use of calcium channel blockers in general or history of use of calcium channel blockers in the treatment of the fissure
8. Signs of other rectal diseases, fistula, infection including severe perianal eczema and tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
Complete healing at week 12 | 12 weeks
  Complete healing of the anal fissure after 12 weeks

SECONDARY OUTCOMES:
Complete healing at week 8 | 8 weeks
  Complete healing of the anal fissure after 8 weeks
Defecation pain at day 3 | 3 days
  Perianal pain at or after defecation at day 3
Defecation pain at day 7 | 7 days
  Perianal pain at or after defecation at day 7
Adverse events | 12 weeks
  Any adverse events recorded during the study period

OTHER OUTCOMES:
Incontinence | 8 and 12 weeks
  Cleveland Clinic incontinence score
Anal resting pressure | 8 and 12 weeks
  Anal resting and maximal pressure measured by anal manometry (Peritron)

CONTACTS AND LOCATIONS:
Overall Officials: Peter-Martin Krarup, MD, Study Chair — Bispebjerg Hospital; Andreas Nordholm-Carstensen, MD, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Department of Surgery P, Aarhus University Hospital, Aarhus
  - Digestive Disease Center, Bispebjerg Hospital, Copenhagen

REFERENCES:
- [Derived] Nordholm-Carstensen A, Perregaard H, Wahlstrom KL, Hagen KB, Hougaard HT, Krarup PM. Treatment of chronic anal fissure: a feasibility study on Levorag(R) Emulgel versus Diltiazem gel 2. Int J Colorectal Dis. 2020 Apr;35(4):615-621. doi: 10.1007/s00384-020-03515-z. Epub 2020 Jan 24. PMID 31980871